CLINICAL TRIAL: NCT04746092
Title: The Capability of Haemato-oncology Patients to Generate Antibodies Against COVID-19 After Infection and Vaccination
Brief Title: The Capability of Haemato-oncology Patients to Generate Antibodies Against COVID-19
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Sponsor
Other Study IDs: 1068-20
Record Dates: First submitted 2021-02-02; First posted 2021-02-09 (Actual); Last update posted 2021-08-16 (Actual); Status verified 2021-02

CONDITIONS: CLL; Multiple Myeloma; Lymphoma
MeSH Terms: conditions — Multiple Myeloma; Lymphoma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The corona pandemic is a continuing global challenge due to Corona Virus 2019 (COVID-19).

The purpose of the study is to evaluate the capability of Haemato-oncology patients to generate antibodies against COVID-19 after infection and vaccination.

DETAILED DESCRIPTION:
In December 2019, a backlog of patients with respiratory disease was identified in Hubei Province, China. The number of infections increased rapidly, and more patients were identified in other provinces in China, and in various countries in the Far East, Europe and the United States. With few exceptions, patients became infected while staying in China. The cause of the disease has been identified as a virus from the corona family - SARS-CoV-2 and the new name given to the disease. (COVID-19) Coronavirus disease The virus belongs to a family of respiratory viruses that often cause mild respiratory illness, however, viruses from this family have also caused epidemics of severe respiratory infections. On March 11, 2020, the World Health Organization declared the corona virus a global pandemic. The average incubation period (from exposure to the onset of clinical symptoms) is 6 days, with a range of 2 to 11 days. Common symptoms of coronary heart disease include: fever, cough, shortness of breath, muscle aches.Some patients develop complications, including pneumonia, respiratory failure, myocarditis and death. Similar to other respiratory viruses, 2019-nCov is transmitted by respiratory droplets. Diagnosis is made by PCR examination from a sample of the upper respiratory tract (pharynx and nose).

In the literature accumulated in recent months suggests that haemato-oncology patients are at increased risk for severe corona disease and mortality. In haemato-oncology patients the recovery process from corona may be prolonged, including a prolonged secretion of the virus compared to a healthy population.

The study population: CLL, Multiple Myeloma or Lymphoma patients as well control group of healthy patients who are vaccinated with COVID-19 in a commercial preparation, regardless of the study.

Serology test between two and three weeks after the second dose of the vaccine to test the effectiveness of the vaccine will be performed as part of the study .During the follow-up period in patients who have developed antibodies to the virus, patients will be offered to repeat the serological test after six months, irrespectively of whether they received a third vaccine within the Israeli standard of care.

All data collected in the study will be typed into Excel and analyzed using SPSS version 21.0. Continuous data will be described using averages and standard deviations, and categorical data will be described using prevalence and percentages.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old
* Patient sex - male and female
* CLL, Lymphoma or Multiple Myeloma patients, in follow up or during an active treatment period, who have recovered from COVID19 (COVID19 recovery defined as the presence of two negative PCR tests), who have been vaccinated against the virus or patients who plan to be vaccinated against COVID19
* Healthy participants who have been vaccinated against the virus as a control group.

Exclusion Criteria:

* Irrelevant

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: CLL, Lymphoma or Multiple Myeloma patients and and their caregivers - healthy participants.
Sampling Method: Non-Probability Sample
Enrollment: 630 (Actual)
Dates: Start 2021-01-06 (Actual); Primary Completion 2022-05-24 (Estimated); Study Completion 2022-05-24 (Estimated)

PRIMARY OUTCOMES:
Capability of Haemato-oncology patients to generate antibodies against COVID-19 after infection and vaccination. | 14 to 21 days counting since second vaccination is initiated.
  Evaluate the capability of Haemato-oncology patients to generate antibodies against COVID-19 after infection and vaccination by using serology tests.

SECONDARY OUTCOMES:
Assess COVID19 morbidity rates | 12-month follow-up as part of routine clinic visits.
  Assess COVID19 morbidity rates in hematologic patients receiving vaccine. patients informs the attending physician in case of diagnosis / infection by COVID 19.
Documentation of the vaccine side effects | 14 to 21 days counting since second vaccination is initiated.
  Documentation of the vaccine side effects among haemato-oncology patients by questioning patients while taking the blood sample.
Comparison of antibody formation to COVID19 between haemato-oncology patients and healthy participants | During the results processing phase about a year and a half from the beginning of the study
  Comparison of antibody formation to COVID19 between haemato-oncology patients and healthy participants by comparing their serology tests.

CONTACTS AND LOCATIONS:
Overall Officials: Yair Herishanu, Prof., Principal Investigator — Tel-Aviv Sourasky Medical Center
Locations (1):
- Tel-Aviv Sourasky Medical Center, Tel Aviv, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Perry C, Luttwak E, Balaban R, Shefer G, Morales MM, Aharon A, Tabib Y, Cohen YC, Benyamini N, Beyar-Katz O, Neaman M, Vitkon R, Keren-Khadmy N, Levin M, Herishanu Y, Avivi I. Efficacy of the BNT162b2 mRNA COVID-19 vaccine in patients with B-cell non-Hodgkin lymphoma. Blood Adv. 2021 Aug 24;5(16):3053-3061. doi: 10.1182/bloodadvances.2021005094. PMID 34387648
- [Derived] Herishanu Y, Avivi I, Aharon A, Shefer G, Levi S, Bronstein Y, Morales M, Ziv T, Shorer Arbel Y, Scarfo L, Joffe E, Perry C, Ghia P. Efficacy of the BNT162b2 mRNA COVID-19 vaccine in patients with chronic lymphocytic leukemia. Blood. 2021 Jun 10;137(23):3165-3173. doi: 10.1182/blood.2021011568. PMID 33861303